CLINICAL TRIAL: NCT05143008
Title: Strategies for Self-Management Around the Reproductive Transition: A Pilot Study
Brief Title: A Pilot Study to Evaluate an Intervention for Gestational Weight Gain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Michele Levine, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO15060569
Record Dates: First submitted 2021-11-18; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Pregnancy Related; Weight Gain; Maternal
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Intervention Model Description: Each participant will be provided with counseling sessions throughout the course of their pregnancy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMART Intervention (Experimental): Counseling sessions will be completed with a toolbox approach so that clinicians can work on topics that are of interest and relevant to each participant. SMART will focus on weight, physical activity, eating and psychosocial issues. Intervention goals will emphasize adherence to healthy behaviors rather than absolute weight goals. Specifically, women will receive consultation about nutritional balance, dietary guidelines for pregnant women and advice to maintain an optimal rate of weight gain according to prepregnancy BMI. Women will use self-monitoring forms to identify and modify cues for unhealthy behaviors. Beliefs about body weight and eating during pregnancy will be addressed and effects of physical activity on body weight, health, and mood will be included.
  Interventions: Behavioral: SMART Intervention

INTERVENTIONS:
Behavioral: SMART Intervention — Counseling sessions will be conducted by research project staff that has, at least, masters level or equivalent degrees. Sessions will occur up to 10 times at their regularly scheduled obstetric appointments and also weekly by phone and text messages. In person sessions will last approximately 20-30 minutes.

SUMMARY:
The purpose of this study is to enable the investigator to conduct proof of concept work related to the feasibility, acceptability, initial efficacy and mechanisms of action (focusing on maternal and infant modifiable factors) for a novel self-management intervention for pregnant women.

DETAILED DESCRIPTION:
This proposed study aims to adapt intervention to address excessive gestational weight gain and psychosocial functioning among a socioeconomically and racially diverse sample of pregnant women .Additionally, data on behavioral mechanisms associated with self-regulatory capacity, such as impulsive control and the ability to delay rewards, that may be linked to self-regulation during pregnancy are needed to support future interventions.

In this study, the investigators will develop and adapt an intervention (Self-Management Around the Reproductive Transition; SMART) that addresses maternal weight, stress, and mood, and document the feasibility, acceptability and initial efficacy of the SMART intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least 14 years of age
* Less than 16 weeks gestation
* English speaking
* Singleton pregnancy
* Receiving care at Magee-Womens Hospital, Latterman family health or other UPMC practices that provide obstetric care

Exclusion Criteria:

* Preexisting diabetes
* Use of medications known to affect weight
* Enrolled in current weight management programming
* History of weight loss surgery
* Women who endorse acute psychiatric symptoms (e.g., suicidality) that warrant immediate care

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2017-02-19 (Actual); Study Completion 2017-02-19 (Actual)

PRIMARY OUTCOMES:
Number of sessions attended among women enrolled in the study | Approximately 9 months
  Number of sessions attended will be calculated for each participant
Number of self-monitoring forms returned | Approximately 9 months
  Number of self-monitoring forms returned will be calculated for each participant
Gestational weight gain | Approximately 9 months
  Gestational weight gain will be calculated for each participant. Weight in pounds will be measured on a calibrated scale while women are in street clothes without shoes.

SECONDARY OUTCOMES:
Depressive symptoms | Approximately 12 months
  The Center for Epidemiological Studies-Depression Scale will be used to assess depressive symptomatology. A total scores is calculated by finding the sum of the 20 items. Total scores range from 0-60, with higher scores reflecting greater depressive symptomatology.
Perceived stress symptoms | Approximately 12 months
  The Perceived Stress Scale will be administered to measure symptoms of perceived stress. The Perceived Stress Scale score is obtained by summing the points awarded to the 10 items and it ranges from 0 to 40. Higher scores indicate greater perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Levine, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No